CLINICAL TRIAL: NCT01167673
Title: A Double Blind Placebo Controlled Cross Over Study for the Use of Coltect (Green Tea, Selenium and Curcumin) in Irritable Bowel Syndrome
Brief Title: The Effect of Coltect (Selenium, Curcumin and Green Tea) on Irritable Bowel Syndrome
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: NAFTALI TIMNA (Other)
Responsible Party: Sponsor-Investigator, NAFTALI TIMNA, MD, Meir Medical Center
Organization: Meir Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: bp004
Record Dates: First submitted 2010-07-21; First posted 2010-07-22 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-06

CONDITIONS: Irritable Bowel Syndrome
Keywords: irritable bowel syndrome; selenium; curcumin; green tea
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- treatment with study drug (Active Comparator): patients receiving study drug for 4 weeks. 3 capsules a day of coltect
  Interventions: Dietary Supplement: coltect
- placebo (Placebo Comparator): patients receiving similar capsules but no active ingredients
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: coltect — green tea 250 mg, selenium 100 micro gram, curcumin 500 mg
  Arms: treatment with study drug
Dietary Supplement: Placebo — placebo
  Arms: placebo

SUMMARY:
Irritable bowel syndrome (IBS) causes many symptoms, including abdominal pain, irregular bowel movements and bloating. It may be caused by loe degree inflammation of the intestine. The ingredients of coltect which contains green tea, selenium, and curcumin have been proven very safe and have anti inflammatory and anti oxidant activity. The aim of the study is to see whether the use of Coltect can improve symptoms in IBS patients.

DETAILED DESCRIPTION:
The etiology of Irritable bowel syndrome is unknown but some evidence suggests it may be caused by a certain degree of inflammation, another theory is that intestinal flora has an influence on IBS. Coltect combines 3 ingredients: green tea, selenium and curcumin, all of which have been shown to have anti inflammatory and anti oxidant activity. the aim of the study is to investigate if use of coltect can improve symptoms in IBS patients

ELIGIBILITY:
Inclusion Criteria:

* IBS as defined by the Rome III criteria
* for those above age 40 a colonoscopy within the last 5 years
* no new treatment in the last 2 weeks
* not receiving any antibiotics in the last 2 weeks

Exclusion Criteria:

* any large abdominal operation (such as colectomy) in the past
* a known disease of the gastrointestinal tract
* any significant debilitating disease such as sever heart failure, un controlled diabetes,

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-04; Primary Completion 2017-12 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
improvement of IBS symptoms and quality of life | 10 weeks
  improvement of IBS symptoms and quality of life (QOL) assessed by IBS and QOL questionaires.

SECONDARY OUTCOMES:
change in bacterial stool flora | 10 weeks
  stool tests to investigate change in intestinal flora during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Timna Naftali, MD, Principal Investigator — Meir MC
Locations (1):
- Gastroenterology institute Meir Hospital, Kfar Saba, Israel